CLINICAL TRIAL: NCT03221946
Title: A Comparative Evaluation of Diclofenac Sodium Transdermal Patch, Oral Diclofenac Sodium With Intramuscular Injections of Diclofenac Sodium in Patients Suffering From Oral Pain: A Randomized Control Trial
Brief Title: A Comparative Evaluation of Diclofenac Sodium Transdermal Patch, Oral Diclofenac Sodium With Intramuscular Injections of Diclofenac Sodium in Patients Suffering From Oral Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, NALLAN CHAITANYA, Clinical Associate Professor, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMVIDS&RC/IEC/OMR/PR 0051-15
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Orofacial Pain
MeSH Terms: conditions — Facial Pain | interventions — Diclofenac; dicloran

STUDY DESIGN:
Intervention Model Description: 3 arms with 3 groups of 30 patients each evaluated for diclofenac sodium oral tablets, transdermal patch and injection of same drug for dental pain disorders
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diclofenac sodium oral (Active Comparator): Group A which included 30 patients of either gender. Dosage drug: Diclofenac sodium Dosage form: Oral medication Frequency: twice daily Dose: 50mg Duration: 2 days
  Interventions: Drug: Diclofenac Sodium
- diclofenac sodium patch (Experimental): Group B which included 30 patients who were prescribed Drug: Diclofenac sodium Dose: 100mg Drug form: transdermal patch to equate the oral dosage of 50mg Duration: for 2 days Frequency: Once daily
  Interventions: Drug: Diclofenac sodium
- Diclofenac sodium injection (Other): Group C which included 30 patients of either gender Drug: diclofenac sodium intra muscular injections Dose: 75mg which was the nearest available dosage to 100 mg availability in India Frequency: once daily Duration: for 2 days
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac Sodium — tablet of 50mg,
  Other Names: Voveran
  Arms: Diclofenac sodium oral
Drug: Diclofenac sodium — Transdermal patch 100 mg
  Other Names: Sparsh
  Arms: diclofenac sodium patch
Drug: Diclofenac — intra muscular injection 100mg
  Other Names: dicloran
  Arms: Diclofenac sodium injection

SUMMARY:
Newer drug delivery systems such as transdermal patches using pain relieving or modifying agents emerged as mainstream treatment protocol for management of pain on the outpatient basis. The administration of Diclofenac 100 mg in transdermal patch in the patients having dental pain due to periapical/periodontal infections was evaluated.

Methods: 90 Patients of either gender, between 18 to 80 years were divided into 3 groups (Group A- oral medication, Group B- transdermal patch, Group C - intra muscular group). Patients at the dental department with pain from periapical/periodontal pathologies were explained about the procedure of analgesia. With written consent, 100 mg diclofenac sodium transdermal patches were prescribed to patients who opted their use in pain control for 2 consecutive days. A Visual Analog Scale was provided for all patients assessing the pain intensity during the study.

DETAILED DESCRIPTION:
Transdermal Patches ensure simple, painless procedure of drug usage even in patients with needle phobia. they are on par with sustainable plasma levels comparable with that of oral medication. With the local drug delivery method, hepatic first pass metabolism is bypassed. Offering increased flexibility in placing and removing the transdermal patch better patient compliance is achieved.

This study was carried out comparing the efficacy of analgesia, occurrence of side effects from the drugs employed and patient compliance during the drug usage with diclofenac sodium trans dermal patch 100 mg, oral supplementation of diclofenac sodium 50 mg given as twice daily medication and intra muscular administration of 75 mg diclofenac sodium once daily for two days in patients having dental pain due to periapical or periodontal pathology.

Material and Methods

A total sample of 90 subjects of either gender, between 18 to 80 years attending Department of Oral Medicine & Radiology with dental pain and who were willing to be part of the study were included and divided randomly into 3 groups based on their preference and priority of the route of administration of the drug. As this was a pilot study, a sample size of 90 was chosen according to recommendations by Isaac and Michael, W. B

The study was cleared by ethical clearance committee with necessary approvals. the subjects were informed thoroughly about the study and could withdraw from the study at their choice when there is no relief of pain with the medication.

The groups included in the study were:

Group A which included 30 patients of either gender who were prescribed tablet Diclofenac sodium 50 mg orally twice daily for 2 days which is the preferred adult dose for dental pain disorders

Group B which included 30 patients who were prescribed Diclofenac sodium 100mg transdermal patch to equate the oral dosage of 50mg that is given twice daily once daily for 2 days ( SPARSH PHARMA). It is a transparent patch that gave sustained release of the drug for 24 hours at the local site applied. A total number of 2 patches were given to each patient one per day. The patches were applied at an hairless area on the left or right shoulders which were subsequently replaced the next day to another area of application in order to avoid contact dermatitis in the area of application.

Group C which included 30 patients of either gender who were given intra muscular injection of 75mg which was the nearest available dosage to 100mg availability in India at deltoid or gluteus muscle once daily for 2 days using sterile and aseptic precautions.

All the subjects were prescribed necessary antibiotics for reduction in peri apical /periodontal infections. The rescue medication tablet chosen was Paracetamol 325 mg, if any of the patients opted for further medication for pain relief. Also, a visual analog scale was provided to all the subjects during their presentation to the hospital for 2 consecutive days for treatment. the scales were obtained in all the subjects individually assessing the intensity of pain after the medication intake during the study period. Team of six doctors evaluated the patients in the study. 2 physicians were assigned the task of data collection from the study participants and assigning them into the group chosen by the patients themselves. 2 physicians had evaluated the patients VAS scores clinically and administered the necessary medication to the patients and rest of the doctors had evaluated the patients at each visit, making a note of inter observer variability. The enquiry of following adverse effects were noted from all 3 groups.

Group A: Rash, Itch, Gastritis

Group B: Rash at the delivery site, adherence of patch

Group C: Pain at injection site, Nerve palsy, Hypersensitivity reactions.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral and dental pain due to pulp and periapical pathology
* patients not allergic to any form of medications in terms of NSAIDs.

Exclusion Criteria:

* Unwilling and unconscious patients
* patients with cellulitis and spreading oral infections
* patients allergic to non steroidal anti inflammatory agents
* patients with kidney and liver diseases
* patients with blood disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Pain Perception scale | 2 days
  Measurement of pain on Visual Analog scale scores in all three groups

SECONDARY OUTCOMES:
Patient compliance - Self reported daily catalog | 2 days
  Self reported by patients themselves on their compliance with oral medication, transdermal patch and intra muscular injection

CONTACTS AND LOCATIONS:
Locations (1):
- Panineeya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No